CLINICAL TRIAL: NCT05681052
Title: Mottling Score and Central Venous Oxygen Saturation in Septic Shock Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Erzincan University (Other)
Responsible Party: Principal Investigator, Nurcan Kutluer Karaca, Asistant Profesor, Erzincan University
Other Study IDs: University of Erzincan
Record Dates: First submitted 2022-12-23; First posted 2023-01-11 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Central Oxygen Saturation; Microcirculation; Mottling Score; Septic Shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Mottling score and central venous oxygen saturation are described as a clinical evaluation of tissue perfusion. This study describes mottling incidence and mottling score in septic shock patients according to central venous oxygen saturation.

DETAILED DESCRIPTION:
This study prospectively analyzed the data of patients admitted to our ICU between October 2022 to December 2022. All septic patients in whom the ScvO2 was measured and mottling scores were evaluated were included. This study enrolled patients aged ≥ 18 years in septic shock. Those excluded have peripheral arterial disease, black skin, cutaneous infection of the lower limbs, pregnancy, and relative refusal. The characteristics of patients were recorded at admission (H0), including demographics (age, sex, body mass index (BMI), admission the Acute Physiology and Chronic Health Evaluation (APACHE II) score, Glasgow Coma Scale (GCS) and sequential organ failure assessment (SOFA) score. Variables such as plasma lactate level, daily urine output, plasma creatinine level, the ratio of arterial oxygen pressure related to inspired oxygen fraction (PaO2/FiO2), hemoglobin level, heart rate, mean arterial pressure, pulsatile saturation in oxygen (SpO2) and body temperature were recorded at H0 and 6 hours after initial resuscitation (H6).

ELIGIBILITY:
Inclusion Criteria:

* patients aged ≥ 18 years in septic shock.

Exclusion Criteria:

* patients having the peripheral arterial disease
* black skin,
* cutaneous infection of the lower limbs
* pregnancy
* relative refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients aged ≥ 18 years in septic shock
Sampling Method: Non-Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-01-21 (Estimated); Study Completion 2023-01-21 (Estimated)

PRIMARY OUTCOMES:
Difference in mottling incidence according to ScvO2 level during a septic shock. | at 0th hour, admission; at 6th hour after initial treatment
Difference in mottling score according to ScvO2 level during a septic shock. | at 0th hour, admission; at 6th hour after initial treatment
  0 score is minimum level, meaning no mottling, meaning better outcome 5 score is maximum level, meaning more mottling, meaning worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Nurcan Kutluer Karaca, Erzincan, Turkey (Türkiye)